CLINICAL TRIAL: NCT06021002
Title: Nasal Immune Challenge Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Akhilesh Jha, Clinical Lecturer in Respiratory Medicine, Cambridge University Hospitals NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A095696
Record Dates: First submitted 2023-08-21; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Innate Inflammatory Response; Asthma; Nasal Allergy
MeSH Terms: conditions — Inflammation; Asthma | interventions — resiquimod; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Single nasal challenge R848 allergic rhinitis (Other)
  Interventions: Drug: R848
- Single nasal challenge R848 healthy (Other)
  Interventions: Drug: R848
- Single nasal challenge saline (Other): Single nasal challenge saline allergic rhinitis and healthy
  Interventions: Drug: Saline
- Repeat nasal challenge R848 allergic rhinitis (Other)
  Interventions: Drug: R848
- Repeat nasal challenge R848 healthy (Other)
  Interventions: Drug: R848
- Repeat nasal challenge saline (Other): Repeat nasal challenge saline allergic rhinitis and healthy
  Interventions: Drug: Saline
- Sample collection only (No Intervention): Sample collection only (no nasal challenge) to optimise laboratory protocols

INTERVENTIONS:
Drug: R848 — Nasal R848 administration
  Arms: Repeat nasal challenge R848 allergic rhinitis; Repeat nasal challenge R848 healthy; Single nasal challenge R848 allergic rhinitis; Single nasal challenge R848 healthy
Drug: Saline — Nasal saline administration
  Arms: Repeat nasal challenge saline; Single nasal challenge saline

SUMMARY:
Respiratory viral infections cause significant illness, especially in vulnerable individuals and is a topic of immense significance during the current COVID-19 global pandemic. Respiratory diseases such as asthma involve inflammation of the airways and viruses are a major cause of asthma attacks. The nose is easier to access than the lungs but has similar cells and is therefore useful to study immune responses throughout the respiratory tract.

Rather than study the effects of a live virus on the immune system, it is possible to give a component or mimic of a virus to simulate an infection in a similar but more straightforward manner, without causing disease.

In this study we will use a nasal spray containing a sterile substance called Resiquimod (also called R848) to mimic a viral infection. Resiquimod does not contain any living organisms and therefore there is no possibility of developing a real infection.

Resiquimod works by binding to receptors in cells that line the inside of the nose (epithelial cells) as well as cells that can fight infection (immune cells). These cells respond to Resiquimod and cause mild inflammation in the nose, similar to a mild cold. We can then take samples to measure this response and investigate how it differs between individuals. This will help us better understand how the human immune system responds to viruses, and which cells and molecules the body uses to defend itself against infection.

DETAILED DESCRIPTION:
Background Acute respiratory viral infections cause significant morbidity, especially in vulnerable individuals and is a topic of immense significance during the current COVID-19 global pandemic. Respiratory diseases such as asthma and chronic obstructive pulmonary disease (COPD) involve inflammation of the airways and viruses are a major cause of exacerbations. Whilst new biological drugs targeting allergic and eosinophilic immune pathways have been developed for allergic asthma, therapeutic options for treating asthma exacerbations remain limited and rely on decades-old blunt tools such as oral corticosteroids. Development of new therapies and vaccines to combat viral respiratory tract infections is slow, partly because of the limited understanding of innate immune responses at the respiratory mucosal site of disease. Detailed characterization of such responses can facilitate biomarker definition for respiratory diseases, providing mechanistic insights and a platform for the testing of novel therapeutics.

Our understanding of the role of innate immunity to infection has recently undergone a paradigm shift as it is now recognized that innate cells (and not just adaptive immune cells) have the capacity to undergo "training" after infection via metabolic changes and epigenetic reprogramming. Pathogens can therefore modulate chromatin structure and the transcriptional programme of innate immune cells, which can result in altered but non-specific responses upon reinfection either with the same or heterologous stimuli. These epigenetic mechanisms may be particularly relevant in understanding how viral triggers (e.g. influenza) can lead to increased susceptibility to bacterial infections and cause pneumonia (e.g. due to streptococcus spp.).

Most studies have focused on peripheral immune cells such as macrophages, but the concept of innate immune training has been extended to long-lived non-immune skin epithelial stem cells, which have the capacity for "inflammatory memory". Allergic inflammatory memory has also recently been established in respiratory progenitor cells. Murine studies have highlighted the potential for structural cells (such as epithelial cells) to have the potential to mount immune responses. However, mechanisms of innate immune "memory" in human respiratory mucosal epithelial and immune cells in response to microbes and pathogen associated molecular patterns (PAMPs) are not well understood despite the respiratory tract being under a constant barrage of infectious stimuli.

Toll-like receptors (TLRs) play a critical role in the initial detection of microbes and PAMPs. TLR7/8 specifically detects RNA viruses such as influenza, rhinovirus, and coronavirus. Airway epithelial and immune cells express TLR7/8 and are therefore vital in mounting the innate immune response to viral infections, as well as helping shape adaptive immunity. Resiquimod (R848) is a single-stranded RNA viral analogue that binds to TLR7/8. When given systemically to treat human hepatitis C infection, it causes cytokine release and a flu-like syndrome. However, R848 has been successfully employed topically as a skin cream for actinic keratosis. TLR7 agonists have been developed for therapeutic use by repeated dose intranasal administration to target allergic inflammation in healthy volunteers and those with allergic rhinitis.

Rationale for current study Intranasal R848 administration has now been established in a human challenge model in healthy volunteers and in those with allergic rhinitis (AR) and allergic rhinitis with asthma (ARwA) by the chief investigator. In total, 44 volunteers have received intranasal R848 at a range of doses; 9 healthy volunteers received 10µg per nostril (n=9) with one person receiving 100µg per nostril (n=1); subsequently 35 volunteers received between 1-2µg per nostril based on weight (0.02µg/kg, healthy n=12, AR n=12, ARwA n=11). This dose was well tolerated by all volunteers with minimal nasal symptoms and no significant change in airflow obstruction (FEV1) in volunteers with asthma. Intranasal R848 was well tolerated systemically with no change in physiological measures or serum inflammatory mediators compared to saline challenge. The study demonstrated that individuals with AR and ARwA have increased nasal mucosal interferon and chemokine responses compared to healthy volunteers. This is coupled with the observation that there is a small and transient reduction in peripheral eosinophil counts at 4 hours and in lymphocyte counts at 24 hours, a finding limited to volunteers with AR and ARwA. This suggests that leukocyte trafficking may be occurring from the peripheral blood to the nasal mucosa. These findings highlight that dysregulated mucosal innate immune responses are likely to be important in determining the clinical outcome of viral triggers.

R848 nasal challenge (up to 2µg per nostril) is therefore a practical, tolerable, and non-invasive method to stimulate and investigate TLR-driven respiratory mucosal innate immune responses in both health and disease.

Defining the cellular basis for TLR-driven innate immunity will help provide mechanistic insights into how these responses differ between individuals, its dysregulation in disease (such as during an asthma exacerbation) and susceptibility to secondary infections. Understanding the epigenetic mechanisms which regulate interferon and chemokine production may help identify the molecular drivers of excessive or dampened inflammation, helping to refine potential therapeutic targets. Given the current COVID-19 pandemic, the clinical translational model utilised in this study allows for a practical and straightforward method to assess the host factors which determine respiratory mucosal innate immunity.

The goal of this project is to utilize an established tolerable human nasal TLR agonist challenge model combined with single-cell transcriptomic and epigenetic techniques to precisely characterize innate immune responses and mechanisms of innate immune training in airway epithelial and immune cells. Samples will be collected from the nasal mucosa and blood before and after saline and R848 challenge. Cell cultures from airway epithelium and blood will also be established to assess the functional impact of R848 on cellular response to repeat stimulation with viral and bacterial ligands. Study populations will include healthy participants and those with allergic rhinitis with/without asthma in order to investigate how in-vivo innate immunity is altered in these populations. Some participants will also undergo repeat nasal challenge to assess mechanisms of innate immune memory in the respiratory tract.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or female aged 18 years and above
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.
* Female participants of child-bearing potential and male participants whose partner is of child-bearing potential must be willing to ensure that they or their partner use effective contraception during the study
* Participant has clinically acceptable laboratory and ECG at enrolment.
* Negative lateral flow or polymerase chain reaction (PCR) test for SARS-CoV-2
* For healthy volunteers:

  * No clinical history of allergic rhinitis, asthma or eczema
  * Negative skin prick tests or specific IgE response to a panel of common aeroallergens: cat, dog, grass pollen, tree pollen, house dust mite, fungal spores
  * Normal blood eosinophil count (< 300 cells/μL)
  * Normal baseline forced expiratory volume (FEV1) i.e. ≥80%
* For volunteers with allergic rhinitis with or without asthma:

  * A clinical history of allergic rhinitis symptoms (sneezing, runny or itchy nose) in response to aeroallergens
  * At least one positive skin-prick test or specific IgE response to a panel of common aeroallergens: cat, dog, grass pollen, tree pollen, house dust mite, fungal spores
  * Pre-bronchodilator FEV1 ≥50% predicted
  * Participants are permitted to have physician-diagnosed mild to moderate asthma which is not poorly controlled as evidenced by an Asthma Control Questionnaire (ACQ-5) score of ≤1.5.
  * If they have asthma, they are permitted to be on inhaled corticosteroid (ICS) and a long-acting beta agonist (LABA), but no other controller medication.
* Have had no other courses of medication including nasal and systemic corticosteroids, whether prescribed or over-the-counter, in the four weeks before first study dose other than mild analgesia, vitamins and mineral supplements or, for females, oral contraceptives.

Exclusion Criteria:

* Recent infections in past 14 days before screening: especially upper respiratory tract illnesses (including colds and influenza), sore throats, sinusitis, infective conjunctivitis.
* Lower respiratory tract infection in past 28 days
* Nasal anatomical defects, precluding use of nasal sampling techniques
* The participant may not enter the study if any of the following apply:

  * Female participants who are pregnant, lactating or planning pregnancy during the study.
  * Respiratory diseases (other than hay fever or asthma where specified)
  * Significant medical history of hepatic, cardiovascular, gastrointestinal, renal, endocrine, infective, haematological, autoimmune, metabolic, rheumatological, neurological, dermatological or neoplastic conditions
  * Extreme obesity (BMI >40)
  * Depression and psychiatric disorders
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks
* Smoking in previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Nasal CXCL10 gene expression baseline vs post-challenge | 24 hours
  Increase in CXCL10 nasal mucosal gene expression at 24 hours after nasal challenge with R848 compared to baseline.

SECONDARY OUTCOMES:
Nasal CXCL10 gene expression between healthy and allergic rhinitis participants | 24 hours
  Difference in CXCL10 nasal mucosal gene expression at 24 hours after R848 challenge between healthy subjects and those with allergic rhinitis.
Average body temperature comparison between first and second nasal R848 challenge | 2 weeks
  Change in participant's temperature between first and second nasal challenge with R848 (as a marker of clinical tolerability).
Nasal CXCL10 AUC between first and second nasal challenge | 2 weeks
  Difference in CXCL10 nasal mucosal protein in nasal mucosal lining fluid over 24 hours expressed as area under curve (AUC) between first and second nasal challenge with R848.
Nasal CXCL10 gene expression saline vs R848 single challenge | 24 hours
  Difference in nasal CXCL10 gene expression after saline and R848 single challenge
Nasal CXCL10 gene expression saline vs R848 repeat challenge | 2 weeks
  Difference in nasal CXCL10 gene expression after saline and R848 repeat challenge

OTHER OUTCOMES:
Blood CXCL10 response to lipopolysaccharide (LPS) | 24 hours
  Difference in CXCL10 after ex-vivo stimulation of blood samples with LPS before and 24 hours after nasal challenge with R848

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jha A, Thwaites RS, Tunstall T, Kon OM, Shattock RJ, Hansel TT, Openshaw PJM. Increased nasal mucosal interferon and CCL13 response to a TLR7/8 agonist in asthma and allergic rhinitis. J Allergy Clin Immunol. 2021 Feb;147(2):694-703.e12. doi: 10.1016/j.jaci.2020.07.012. Epub 2020 Jul 24. PMID 32717253

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT06021002/Prot_SAP_000.pdf